CLINICAL TRIAL: NCT03861143
Title: A Randomized , Placebo-Controlled, Double-Blind, Multicenter Study to Evaluate Efficacy and Safety of Oral BT-11 in Ulcerative Colitis
Brief Title: Efficacy and Safety of Oral BT-11 in Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NImmune Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BT-11-201
Record Dates: First submitted 2019-02-27; First posted 2019-03-04 (Actual); Results first posted 2022-11-03 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Intervention Model Description: This is a phase 2 randomized, placebo-controlled, double-blind, parallel-group multicenter study with an optional open label extension (OLE) period. The purpose of this study is to evaluate the efficacy and safety of oral BT-11 compared to placebo in subjects with UC. This study includes 3 periods: induction, maintenance, and an optional OLE period.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- BT-11 low-dose (440 mg) (Experimental): Oral, once daily tablet
  Interventions: Drug: BT-11 (440 mg)
- BT-11 high-dose (880 mg) (Experimental): Oral, once daily tablet
  Interventions: Drug: BT-11 (880 mg)
- Placebo (Placebo Comparator): Oral, once daily tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BT-11 (440 mg) — Oral, once daily tablet
  Arms: BT-11 low-dose (440 mg)
Drug: BT-11 (880 mg) — Oral, once daily tablet
  Arms: BT-11 high-dose (880 mg)
Drug: Placebo — Oral, once daily tablet
  Arms: Placebo

SUMMARY:
This is a phase 2 randomized, placebo-controlled, double-blind, parallel-group multicenter study with an optional open-label extension (OLE) period. The purpose of this study is to evaluate the efficacy and safety of oral BT-11 compared to placebo in subjects with UC. This study includes 3 periods: induction, maintenance, and an optional OLE period.

ELIGIBILITY:
Key Inclusion Criteria:

1. . Male and female subjects aged 18 to 75 years, inclusive.
2. . Diagnosis of UC for at least 3 months prior to screening.
3. . UC, as defined by a total Mayo Score of 4 to 10 inclusive at baseline with a MES 2 (confirmed by central reader).
4. . Able to participate fully in all aspects of this clinical trial.
5. . Written informed consent must be obtained and documented.

Key Exclusion Criteria:

1. . A diagnosis of CD, indeterminate colitis, or presence or history of the fistula with CD.
2. . Modified Truelove and Witts criteria (2: 6 bloody stools per day and one or more of the following: pulse > 90 bpm, temperature > 37.8°C, hemoglobin < 10.5 g/dl, or hs-CRP > 30 mg/I).
3. . Disease activity limited to distal 15 cm (proctitis).
4. . Treatment with an immunosuppressant (azathioprine, 6- mercaptopurine [6-MP]) within 25 days prior to randomization.
5. . Unable to attend study visits or comply with procedures.
6. . Concurrent participation in any other interventional study.
7. . Prior enrollment in the current study and had received study treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2019-08-14 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2021-06-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (9):
  - Axis Clinical Trials, Los Angeles, California
  - Ventura Clinical Trials, Ventura, California
  - Clinical Research of California, Walnut Creek, California
  - Medycal Research Inc., Brooksville, Florida
  - Invesclinic.U.S,LLC.FL, Fort Lauderdale, Florida
  - I.H.S Health LLC, Kissimmee, Florida
  - Smart Medical Research, Richmond Hill, New York
  - Invesclinic.U.S,LLC., McAllen, Texas
  - Texas Gastroenterology Associates, Spring, Texas
- Bosnia and Herzegovina (2):
  - Polyclinic and Daily hospital "Dr Al Tawil", Sarajevo, Federation BiH
  - Cantonal Hospital Zenica, Gastroenterology, Zenica
- Polyclinic Duvnjak, Zagreb, Croatia
- Poland (2):
  - RIVERM E D Sp. zo.o., Poznan, Greater Poland Voivodeship
  - Centrum Badan Klinicznych PI-House Sp. z o.o., Gdansk, Pomeranian Voivodeship
- Ukraine (2):
  - Municipal Non-profit Enterprise "City Outpatient Clinic No 9 of Kharkiv City Council, Surgery department, Kharkiv, Kharkiv
  - Multidisciplinary Medical Center of Odesa National Medical University, First Surgery Department ,Odesa National Medical University , Chair of General and Military Surgeon, Odesa

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BT-11 Low-dose (440 mg) | BT-11 High-dose (880 mg) | Placebo
Started | 66 | 66 | 66
Completed | 62 | 59 | 58
Not Completed | 4 | 7 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BT-11 Low-dose (440 mg) | BT-11 High-dose (880 mg) | Placebo | Total
Number analyzed (Participants) | 66 | 66 | 66 | 198
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.1 (14.9) | 43.3 (14.9) | 43.3 (14.5) | 43.2 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 22 | 31 | 93
  Male | 26 | 44 | 35 | 105
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 2 | 3
  White | 65 | 65 | 64 | 194
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Clinical Remission
Description: Clinical remission rate at Week 12, defined using the 3-component modified Mayo Score as a rectal bleeding subscore of 0, a stool frequency subscore of 0 or 1, and an endoscopic subscore of 0 or 1.
Time Frame: Week 12
Population: ITT
Measure: Number; unit: percentage of participants
Arm/Group | BT-11 Low-dose (440 mg) | BT-11 High-dose (880 mg) | Placebo
Number analyzed (Participants) | 66 | 66 | 66
percentage of participants | 30.3 | 31.8 | 22.7

ADVERSE EVENTS:
Time Frame: 15 months
Arm/Group | BT-11 Low-dose (440 mg) | BT-11 High-dose (880 mg) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/66 | 0/66
Serious Adverse Events (participants affected / at risk) | 2/66 | 3/66 | 3/66
Other Adverse Events (participants affected / at risk) | 23/66 | 29/66 | 27/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BT-11 Low-dose (440 mg) (N=66) | BT-11 High-dose (880 mg) (N=66) | Placebo (N=66)
Colitis Ulcerative (Gastrointestinal disorders) | 0 | 1 | 1
Proctitis (Gastrointestinal disorders) | 1 | 0 | 0
Amoebiasis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1
Pneumonia Viral (Infections and infestations) | 0 | 0 | 1
Foot Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Coronavirus Test Positive (Investigations) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BT-11 Low-dose (440 mg) (N=66) | BT-11 High-dose (880 mg) (N=66) | Placebo (N=66)
Anemia (Blood and lymphatic system disorders) | 2 | 5 | 0
Colitis Ulcerative (Gastrointestinal disorders) | 10 | 8 | 6
Diarrhea (Gastrointestinal disorders) | 3 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 3 | 0
Corona Virus Infection (Infections and infestations) | 1 | 1 | 4
Blood Creatine Phosphokinase Increased (Investigations) | 1 | 3 | 0
Headache (Nervous system disorders) | 0 | 1 | 3
Other (General disorders) | 6 | 8 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-03): https://cdn.clinicaltrials.gov/large-docs/43/NCT03861143/Prot_SAP_002.pdf